CLINICAL TRIAL: NCT03079609
Title: The Search for Viral and Bacterial Etiology of Varicocele
Acronym: ViBaVa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ViBaVa
Record Dates: First submitted 2017-02-08; First posted 2017-03-14 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Varicocele; Viral Infection; Bacterial Infections; Sonic Hedgehog Expression; VEGF Expression
MeSH Terms: conditions — Varicocele; Virus Diseases; Bacterial Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microsurgery urology (Experimental): 20 patients with varicocele (grade II or III) undergoing subinguinal microsurgery varicocelectomy due to infertility and/or pain in the scrotum.
  Interventions: Procedure: subinguinal microscopic varicocelectomy
- open general surgery (Active Comparator): 20 patients (without varicocele) undergoing open hernia repair.
  Interventions: Procedure: open hernia repair

INTERVENTIONS:
Procedure: subinguinal microscopic varicocelectomy — During the procedure approximately 1cm long fragment of varicose vein will be taken for further investigation.
  Arms: microsurgery urology
Procedure: open hernia repair — During the procedure approximately 1cm long fragment of spermatic cord vein will be taken for further investigation.
  Arms: open general surgery

SUMMARY:
This study is to answer the question is there any relationship between viral ( HSV 1 , HSV 2 , HPV 6/11, CMV, HHV 6 , HHV 8, BKV) or bacterial (Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia, Fusobacterium nucleatum) infection and occurrence of varicocele in men.

ELIGIBILITY:
Inclusion Criteria:

* in experimental arm - varicocele grade II or III and infertility and/or pain

Exclusion Criteria:

* in control arm: presence of varicocele in ultrasound before surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Level of presence od viral or bacterial infection, level of expression of SHH and VEGF in varicose vein wall. . | one year after finishing recruitment
  Qualitative and quantitive analysis (presence and concentration - µl or U/µl in two different laboratory tests.) to detect genetic material (DNA, mRNA) of bacteria/viruses will be performed. The outcomes from both gropus will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Dobroński, MD PhD, Study Chair — Chair and Department of Urology Warsaw Medical University
Locations (1):
- Chair and Department of Urology Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Iafrate M, Galfano A, Macchi V, Ejituru E, Sarasin G, Porzionato A, Novara G, De Caro R, Artibani W, Ficarra V. Varicocele is associated with an increase of connective tissue of the pampiniform plexus vein wall. World J Urol. 2009 Jun;27(3):363-9. doi: 10.1007/s00345-008-0352-2. Epub 2008 Nov 22. PMID 19030866
- [Background] Lee JD, Jeng SY, Lee TH. Bcl-2 overexpression in the internal spermatic vein of patients with varicocele. J Formos Med Assoc. 2007 Apr;106(4):308-12. doi: 10.1016/S0929-6646(09)60257-6. PMID 17475608
- [Background] Wang SH, Yang WK, Lee JD. Increased expression of the sonic hedgehog and vascular endothelial growth factor with co-localization in varicocele veins. Phlebology. 2017 Mar;32(2):115-119. doi: 10.1177/0268355515627717. Epub 2016 Jul 9. PMID 26867642
- [Background] Petrovic I, Milivojevic M, Popovic J, Schwirtlich M, Rankovic B, Stevanovic M. SOX18 Is a Novel Target Gene of Hedgehog Signaling in Cervical Carcinoma Cell Lines. PLoS One. 2015 Nov 20;10(11):e0143591. doi: 10.1371/journal.pone.0143591. eCollection 2015. PMID 26588701
- [Background] Hwang J, Kang MH, Yoo YA, Quan YH, Kim HK, Oh SC, Choi YH. The effects of sonic hedgehog signaling pathway components on non-small-cell lung cancer progression and clinical outcome. World J Surg Oncol. 2014 Aug 21;12:268. doi: 10.1186/1477-7819-12-268. PMID 25141859
- [Background] Paulis L, Fauconnier J, Cazorla O, Thireau J, Soleti R, Vidal B, Ouille A, Bartholome M, Bideaux P, Roubille F, Le Guennec JY, Andriantsitohaina R, Martinez MC, Lacampagne A. Activation of Sonic hedgehog signaling in ventricular cardiomyocytes exerts cardioprotection against ischemia reperfusion injuries. Sci Rep. 2015 Jan 23;5:7983. doi: 10.1038/srep07983. PMID 25613906
- [Background] Ai QY, Tian H, Ma L, Miao NZ, Huo YW, Wang HX, Wang LR, Qiu SD, Zhang QY. [Experimental varicocele affects VEGF and Flt-1 protein expressions in the testis and epididymis of adolescent rats]. Zhonghua Nan Ke Xue. 2009 Jun;15(6):488-92. Chinese. PMID 19593986
- [Background] Tek M, Cayan S, Yilmaz N, Oguz I, Erdem E, Akbay E. The effect of vascular endothelial growth factor on spermatogenesis and apoptosis in experimentally varicocele-induced adolescent rats. Fertil Steril. 2009 May;91(5 Suppl):2247-52. doi: 10.1016/j.fertnstert.2008.06.008. Epub 2008 Aug 12. PMID 18701100
- [Background] Kilinc F, Kayaselcuk F, Aygun C, Guvel S, Egilmez T, Ozkardes H. Experimental varicocele induces hypoxia inducible factor-1alpha, vascular endothelial growth factor expression and angiogenesis in the rat testis. J Urol. 2004 Sep;172(3):1188-91. doi: 10.1097/01.ju.0000135455.97627.15. PMID 15311067